CLINICAL TRIAL: NCT02507258
Title: Post Market Clinical Follow-Up Study Protocol for PROFEMUR® Am Femoral Components and PROCOTYL® O HA Coated Acetabular Components
Brief Title: PMCF Study for PROFEMUR® Am Femoral Components and PROCOTYL® O HA Coated Acetabular Components
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision to not renew CE mark on product. Therefore study not needed.
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002K
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Joint Disease
Keywords: osteoarthritis; avascular necrosis; correction of functional deformity; painful hip dysplasia; protrusio acetabuli; rheumatoid arthritis; ankylosis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PROFEMUR® Am Femoral Stem: Single study group previously implanted with a primary PROFEMUR® Am Femoral Stem and PROCOTYL® O HA Coated Acetabular Component
  Interventions: Device: PROFEMUR® Am Femoral Stem w/ PROCOTYL® O Shell

INTERVENTIONS:
Device: PROFEMUR® Am Femoral Stem w/ PROCOTYL® O Shell — PROFEMUR® Am cementless stems with PROCOTYL® O HA Coated Acetabular Component

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of its total hip arthroplasty (THA) and resurfacing components marketed in the European Union (EU). These types of studies are required by regulatory authorities for all THA and resurfacing devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in the EU. This study has been designed in accordance with the medial device directives (MEDDEV) 2.12/2 rev 2.

ELIGIBILITY:
Inclusion Criteria:

Subject has undergone primary THA for any of the following:

* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, or painful hip dysplasia;
* Inflammatory degenerative joint disease such as rheumatoid arthritis; or
* Correction of functional deformity
* Subject is implanted with the specified combination of components
* Subject is willing and able to complete required study visits or assessments

Exclusion Criteria:

* Subjects skeletally immature (less than 21 years of age) at time of primary THA surgery
* Subjects implanted with non-MPO components (femoral stem, femoral head, acetabular liners) in the enrolled THA
* Subjects currently enrolled in another clinical study which could affect the endpoints of this protocol
* Subjects unwilling to sign the Informed Consent document
* Subjects with substance abuse issues
* Subjects who are incarcerated or having pending incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been previously implanted with a PROFEMUR® Am Femoral Stem and PROCOTYL® O HA-Coated Acetabular Component
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary objective of this study is to estimate survivorship using Kaplan Meier analysis of all components at specified intervals out to 10 years follow-up. Measured by capturing date of revision or removal of the device.

SECONDARY OUTCOMES:
Patient functional outcomes (hip specific) | Early (2-5 yrs), Midterm (5-7 yrs), and Long-term (10 yrs + 3 mos) beginning with first available follow-up interval
  To characterize total functional scores, as assessed by Oxford Hip and EQ-5D-3L scores

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Giordano, MD, Principal Investigator — Hopital Joseph Ducuing
Locations (1):
- Hopital Joseph Ducuing, Toulouse, France

IPD SHARING:
Plan to Share IPD: No